CLINICAL TRIAL: NCT02288286
Title: Safety and Immunogenicity of Freeze-dried Rabies Vaccine（MRC-5 Cell) in Chinese Humans From 10-60 Years Old
Brief Title: Safety and Immunogenicity of Freeze-dried Rabies Vaccine（MRC-5 Cell) in Chinese Humans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Center for Disease Control and Prevention (Other Government)
Collaborators: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BJCDCP-11
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2014-11

CONDITIONS: Safety, Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 2.5IU/ml in humans aged 10-20 years old (Experimental): freeze-dried rabies vaccines(MRC-5 cell) of 2.5IU/ml in 200 humans aged 10-20 years old on days 0,3,7,14,28
  Interventions: Biological: 2.5IU/ml rabies vaccine(MRC-5 cell) in humans aged 10-20 years old
- 2.5IU/ml in humans aged 21-50 (Experimental): freeze-dried rabies vaccines(MRC-5 cell) of 2.5IU/ml in 200 humans aged 21-50 years old on days 0,3,7,14,28
  Interventions: Biological: 2.5IU/ml rabies vaccine(MRC-5 cell) in humans aged 21-50 years old
- 2.5IU/ml in humans aged 51-60 (Experimental): freeze-dried rabies vaccines(MRC-5 cell) of 2.5IU/ml in 200 humans aged 51-60 years old on days 0,3,7,14,28
  Interventions: Biological: 2.5IU/ml rabies vaccine(MRC-5 cell) in humans aged 51-60 years old
- 2.5IU/ml in humans(from 10-20 years old) (Placebo Comparator): freeze-dried rabies vaccines(vero cell) of 2.5IU/ml in 200 humans aged 10-20 years old on days 0,3,7,14,28
  Interventions: Biological: 2.5IU/ml rabies vaccine(vero cell) in humans aged 10-20 years old
- 2.5IU/ml in humans(from 21-50 years old) (Placebo Comparator): freeze-dried rabies vaccines(vero cell) of 2.5IU/ml in 200 humans aged 21-50 years old on days 0,3,7,14,28
  Interventions: Biological: 2.5IU/ml rabies vaccine(vero cell) in humans aged 21-50 years old
- 2.5IU/ml in humans(from 51-60 years old) (Placebo Comparator): freeze-dried rabies vaccines(vero cell) of 2.5IU/ml in 200 humans aged 51-60 years old on days 0,3,7,14,28
  Interventions: Biological: 2.5IU/ml rabies vaccine(vero cell) in humans aged 51-60 years old

INTERVENTIONS:
Biological: 2.5IU/ml rabies vaccine(MRC-5 cell) in humans aged 10-20 years old — freeze-dried rabies vaccine(MRC-5 cell) of 2.5IU/ml, 5 doses, 4 weeks interval
  Arms: 2.5IU/ml in humans aged 10-20 years old
Biological: 2.5IU/ml rabies vaccine(MRC-5 cell) in humans aged 21-50 years old — freeze-dried rabies vaccine(MRC-5 cell) of 2.5IU/ml, 5 doses, 4 weeks interval
  Arms: 2.5IU/ml in humans aged 21-50
Biological: 2.5IU/ml rabies vaccine(MRC-5 cell) in humans aged 51-60 years old — freeze-dried rabies vaccine(MRC-5 cell) of 2.5IU/ml, 5 doses, 4 weeks interval
  Arms: 2.5IU/ml in humans aged 51-60
Biological: 2.5IU/ml rabies vaccine(vero cell) in humans aged 10-20 years old — freeze-dried rabies vaccine(vero cell) of 2.5IU/ml, 5 doses, 4 weeks interval
  Arms: 2.5IU/ml in humans(from 10-20 years old)
Biological: 2.5IU/ml rabies vaccine(vero cell) in humans aged 21-50 years old — freeze-dried rabies vaccine(vero cell) of 2.5IU/ml, 5 doses, 4 weeks interval
  Arms: 2.5IU/ml in humans(from 21-50 years old)
Biological: 2.5IU/ml rabies vaccine(vero cell) in humans aged 51-60 years old — freeze-dried rabies vaccine(vero cell) of 2.5IU/ml, 5 doses, 4 weeks interval
  Arms: 2.5IU/ml in humans(from 51-60 years old)

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of freeze-dried rabies vaccine (MRC-5 cells)in different age health human populations, according to the traditional Essen methods (1-1-1-1-1) vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 10-60 years old healthy people with normal intelligence
* Obtain informed consent from the participants or their guardians, and signed informed consent
* The participants or their guardians can comply with the requirements of clinical trial scheme
* The axillary temperature is 37.0 ℃ or less

Exclusion Criteria:

* participants who vaccinated with rabies vaccine before
* participants who used anti-rabies passive immunization agents
* participants who were Suspect or have a history of injury which is hurted by warm-blooded mammals
* Female who was pregnant, or in the lactation period, or have Pregnant plans in the clinical trial.
* participants who have allergy history, especially those who are allergic to neomycin,or had serious adverse reactions ever, Such as allergies, hives, difficulty breathing, angioneurotic edema, or abdominal pain and so on.
* participants who had been diagnosed or suspected to have immunodeficiency or Autoimmune diseases,or have Immune system disorders.
* participants who have Thyroidectomy History,or had been treated because of Thyroid disease in the past year.
* participants who had abnormal clotting which is diagnosed by doctor(such as clotting factor deficiency, coagulation disorders, platelet abnormalities),or who had coagulopathy.
* Participants who had history of epilepsy, seizures or convulsions ,or family history of mental illness.
* Participants who is asplenia, or functional asplenia, and asplenia or splenic resection under any circumstances.
* Participants who had immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids in the past six months. (It does not include Corticosteroid spray treatment Of allergic rhinitis, Surface treatment with corticosteroids because of acute uncomplicated dermatitis)
* Participants who had Received blood products in the past 3 months
* Participants who had Received other investigational drug in the past one month.
* Participants who had received Live attenuated vaccine 14 days before the clinical trial.
* Participants who had received Subunit vaccines and inactivated vaccines 7days before the clinical trial.
* Participants who was having the prevent or the treatment of Antituberculosis.
* Participants who had fever 3 days before receving the Vaccine.( Axillary temperature is above 38℃)
* Participants who was suffering from severe chronic.( Such as Down's syndrome, diabetes, sickle cell anemia or neurological disorder, Guillain-Barre syndrome);
* Participants who was diagnosed or suspected to be suffering from some disease, such as Respiratory diseases, acute infection, Chronic of active stage，Cardiovascular Disease, Severe hypertension, Skin disease ,or the mother or her children was HIV-infected, besides the participants were during the Treatment period of malignant tumors,.
* According to the researchers, there are other factors that are not suitable for Participants to join the clinical trial.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of freeze-dried rabies vaccine(MRC-5 cell) in chinese humans | within the first 4 weeks after the first vaccination
  Adverse reactions associated with vaccine

SECONDARY OUTCOMES:
Evaluate the immunogenicity of freeze-dried rabies vaccine(MRC-5 cell) in chinese humans | within the first 4 weeks after the first vaccination
  Examination of the value of IgE antibody